CLINICAL TRIAL: NCT01620008
Title: Effects of Placental Transfusion on Early Brain Development
Brief Title: Delayed Cord Clamping and Infant Brain Study
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Brown University (Other)
Responsible Party: Principal Investigator, Judith S Mercer, Principal Investigator, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mercer-9329
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Iron Deficiency
Keywords: cord clamping (delayed or immediate); Myelin content; Ferritin
MeSH Terms: conditions — Iron Deficiencies | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: randomized trial (with a preference arm)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Cord Clamping (ICC) (No Intervention): The infant will be placed on the maternal abdomen and the umbilical cord will be clamped immediately after birth (routine care).
- Delayed Cord Clamping (DCC) (Experimental): At birth, infants will be placed on the maternal abdomen and the cord clamping will be delayed for 5 minutes. If the provider is unable to delay the cord clamping, the cord will be milked 5 times.
  Interventions: Procedure: Delayed Cord Clamping

INTERVENTIONS:
Procedure: Delayed Cord Clamping — At birth, the infant will be placed on the maternal abdomen and the umbilical will either be cut immediately or after a 5 minute delay.
  Other Names: delayed umbilical cord clamping
  Arms: Delayed Cord Clamping (DCC)

SUMMARY:
The purpose of this study is to determine if delaying cord clamping at the birth of term infants effects the early brain development (myelin deposition)as determined by quantitative MRI at 4 and 10 months and developmental testing at 4, 10 and 24 months. This study will help to establish a scientific basis for the timing of cord clamping with reference to brain development.

DETAILED DESCRIPTION:
The current obstetrical practice at birth in the United States is that the umbilical cord of the infant is clamped immediately. When immediate clamping occurs, 20 to 40% of the fetal-placental blood volume is left behind in the placenta. This blood contains enough iron-rich red blood cells to meet the infant's iron needs for the first 4 to 6 months of life. Delaying cord clamping has been shown to increase early iron stores without contributing to adverse outcomes. Early iron sufficiency is essential for long term neurologic health. Iron deficiency in infancy adversely affects cognitive, motor, socio-emotional, and behavioral development. Human and animal studies have shown that inadequate iron stores in early infancy have an irreversible negative impact on the developing brain with deficits persisting even after iron levels have been restored by iron supplementation. Iron is an essential component of myelination which is critical for normal brain development and function. Myelination, which peaks during the first year of life, establishes and maintains efficient communication between the discrete regions of the brain. Abnormal myelination underlies a variety of childhood developmental disorders including conditions such as autism.

The gap is that the effect of increased iron stores from delayed cord clamping on myelination and neurodevelopment during early childhood is unknown. Our hypothesis is that placental transfusion affects myelination and early childhood development in the following ways: 1) placental transfusions lead to increased blood volume (BV) and red cell volume (RCV) at birth; 2) increased RCV results in more available iron for early body iron stores; 3) increased body iron stores provide essential iron supply for optimal myelination; 4) optimal myelination results in improved developmental and cognitive performance. We propose a randomized controlled longitudinal (birth to 24 months) trial of 128 infants to measure the effect of placental transfusion on the structure and function of the developing brain. We will use a non-invasive neuroimaging technique to measure myelin acquisition over time and to correlate the findings with iron stores and developmental outcomes. Enrolled women will be randomized at birth to the immediate cord clamping group or the delayed cord clamping group. We will assess infants for iron sufficiency and myelin deposition at 4 and 10 months and evaluate developmental outcomes at 4, 10, and 24 months. This study will help to establish a scientific basis for the timing of cord clamping with reference to brain development. The innovation of this study is in the simplicity of delaying cord clamping combined with the use of a new method of MRI that can quantify myelin deposition. This low-tech change in a clinical practice has the potential to reduce iron deficiency and improve developmental outcomes. If delayed cord clamping demonstrates protective effects for optimal development, changing practice will translate into a large cost savings improving lifetime productivity beneficial to society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* women in the third trimester with:
* singleton pregnancy
* planning to breastfeed for six months
* English speaking
* planning vaginal birth

Exclusion Criteria:

* major medical or obstetrical complications
* Intrauterine growth restriction
* chorioamnionitis
* familial learning disability
* major psychiatric or depressive illness
* fetal congenital anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Brain Myelin Volume | 4 months of age
  At 4 months of age, term infants exposed to delayed cord clamping will have greater myelin content when compared to infants exposed to immediate cord clamping

SECONDARY OUTCOMES:
Ferritin levels | 4 months of age
  Term infants exposed to delayed cord clamping will have higher ferritin levels when compared to infants with immediate cord clamping.

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, CNM, Principal Investigator — Women & Infants Hospital of Rhode Island, University of Rhode Island; Debra A Erickson-Owens, PhD, CNM, Principal Investigator — University of Rhode Island; Women & Infants Hospital of Rhode Island; Sean C. Deoni, PhD, Principal Investigator — Brown University
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Mercer JS, Erickson-Owens DA. Rethinking placental transfusion and cord clamping issues. J Perinat Neonatal Nurs. 2012 Jul-Sep;26(3):202-17; quiz 218-9. doi: 10.1097/JPN.0b013e31825d2d9a. PMID 22843002
- [Background] Mercer JS, Erickson-Owens DA. Is it time to rethink cord management when resuscitation is needed? J Midwifery Womens Health. 2014 Nov-Dec;59(6):635-644. doi: 10.1111/jmwh.12206. Epub 2014 Oct 8. PMID 25297530
- [Derived] Xodo S, Xodo L, Baccarini G, Driul L, Londero AP. Does Delayed Cord Clamping Improve Long-Term (>/=4 Months) Neurodevelopment in Term Babies? A Systematic Review and a Meta-Analysis of Randomized Clinical Trials. Front Pediatr. 2021 Apr 12;9:651410. doi: 10.3389/fped.2021.651410. eCollection 2021. PMID 33912524
- [Derived] Mercer JS, Erickson-Owens DA, Deoni SCL, Dean DC 3rd, Collins J, Parker AB, Wang M, Joelson S, Mercer EN, Padbury JF. Effects of Delayed Cord Clamping on 4-Month Ferritin Levels, Brain Myelin Content, and Neurodevelopment: A Randomized Controlled Trial. J Pediatr. 2018 Dec;203:266-272.e2. doi: 10.1016/j.jpeds.2018.06.006. Epub 2018 Jul 6. PMID 30473033